CLINICAL TRIAL: NCT03259178
Title: Correlation Between Changes in Measures of the Visual System and Changes in Concussion-associated Symptoms
Status: Terminated | Type: Observational
Why Stopped: We were unable to recruit patients because the clinician doing the testing was no longer available between Sep 15 2017 and Mar 1 2018.
Sponsor: McGill University (Other)
Collaborators: Institut National du Sport du Quebec (Unknown); Apexk (Unknown)
Responsible Party: Principal Investigator, Ian Shrier, Principle investigator, McGill University
Other Study IDs: ConBVT
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Concussion; Syndrome
Keywords: Binocular vision test
MeSH Terms: conditions — Brain Concussion; Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sports-related concussion affect 1.6 to 3.8 million people each year in the United States. Despite increased media attention and awareness campaigns, the exact number is difficult to determine due to underreporting by athletes. The types of symptoms experienced with a concussion depend on the area of the brain that was affected. The most frequent symptoms include: headaches, cognitive difficulties, dizziness, neck pain, visual disturbances, difficulty sleeping, and fatigue.

Despite the availability of many treatment options, some patients continue to experience many symptoms - such as headaches, dizziness, visual disturbances, balance problems, sensitivity to light, and difficulties concentrating - that negatively affect school, work, and quality of life for long periods of time. All of these symptoms are similarly experienced by individuals with visual dysfunctions, such as the inability of the eyes to move together. This finding has led some to recommend a visual component in concussion management. Therefore, the purpose of this study is to determine whether changes in the results of 7 binocular vision tests (BVT) over time in patients with concussion correlate with changes in concussion symptoms. The investigators will measure 46 concussion patients aged 18 to 30 years with each of these tests and assess their concussion symptoms on up to four separate visits, which depend on when the patient's symptoms improve.

The tests the investigators will evaluate measure: 3D vision, uniform movement of the eyes, ability of the eyes to adapt to a target moving towards and/or away from the eyes, quick movements of the eyes, natural alignment of the eyes, and double vision as a target is moved towards the eyes. In addition, concussion symptoms will be measured by a standardized concussion questionnaire (SCAT3) at each visit.

The results of each BVT will be entered into a statistical model with the participant's concussion symptom score to determine if there is an association between the change in symptoms and the change in the results of the tests.

DETAILED DESCRIPTION:
Sports-related concussion affect 1.6 to 3.8 million people each year in the United States. Despite increased media attention and awareness campaigns, the exact incidence is difficult to determine due to underreporting by athletes. Concussion is defined as a set of pathological reactions leading to direct damage of the brain, which may occur from a direct or indirect blow to the head. The types of symptoms experienced depend on the area of the brain that was affected. The most frequent symptoms include: headaches, cognitive difficulties, dizziness, neck pain, visual disturbances, difficulty sleeping, and fatigue.

Despite the availability of many treatment options such as neurological and psychological tests, some patients continue to experience many symptoms - such as headaches, dizziness, visual disturbances, balance problems, sensitivity to light, and difficulties concentrating - that negatively affect school, work, and quality of life for long periods of time. All of these symptoms are similarly experienced by individuals with visual dysfunctions such as dysfunctions of binocular function or convergence insufficiency. This finding has led some to recommend a visual component in concussion management. Therefore, the purpose of this study is to determine if changes in the results of 7 binocular vision tests (BVT) over time in patients with concussion correlate with changes in concussion symptoms.

The investigators will measure 46 concussion patients with each of these tests and the SCAT3 on up to 4 separate milestone time points as described below:

* M1 = baseline; as soon as possible after recruitment
* M2 = when participants qualitatively feel that their concussion symptoms have "significantly improved"
* M3 = when participants are symptom-free at with activity for 1 week, or at 3 months post-enrolment in the study, whichever comes first. This milestone will also be the last measurement and mark the end of their participation.
* M* = Participants who do not have significant improvement (i.e. M2) within 2 weeks of baseline testing will also be tested at the 2-week mark. They will still be tested at both M2 and M3.

Demographic information relevant to the study will be collected in order to appropriately describe the population and evaluate the potential effect modification of these factors on the observed correlations. Demographic variables to be recorded include: age, sex, highest level of education achieved, the use of corrective lenses for vision problems, occupation, any relevant past medical history (i.e. migraines, vision problems, medication, etc.), the main sports activity the athlete is involved in, and the last of activities that the athlete will be returning to after healing, with an emphasis on high risk activities for concussions. Furthermore, information relevant to the concussion event will be recorded to characterize the injury. This includes information regarding the accident resulting in concussion, activity at the time of injury, and the mechanism of injury (the presence or absence of head contact is important).

Participants will complete the symptom portion (section 3) of the validated SCAT3 form that is part of the accepted standard for management of concussion. The symptoms listed are: headache, "pressure in head", neck pain, nausea or vomiting, dizziness, blurred vision, balance problems, sensitivity to light or noise, "feeling slowed down", feeling like "in a fog", "don't feel right", difficulty concentrating, difficulty remembering, fatigue or low energy, confusion, drowsiness, trouble falling asleep, more emotional, irritability, sadness, nervous or anxious. Symptoms are scored on a scale of 0 (none) to 6 (severe). The overall symptom score is the sum of all individual symptom scores.

The investigators will include an additional seven questions about symptoms - that are asked by some clinicians: "Symptoms worse with physical activity", "Symptoms worse with mental activity", "Motion sickness", "Discomfort while reading", "Discomfort while using a computer", "Double vision", "Pain behind your eyes". Each symptom is again scored between 0 (none) to 6 (severe).

BVTs will be examined, which differ from optometry tests in that they use more advanced equipment which can measure very small deviations in several domains of the visual system. These BVT measure various elements of the visual system and will be described in detail below:

1. Gross stereoscopic acuity: (range 0 - 15 arc seconds) Our binocular vision allows us to see in three dimensions (3D), or more simply, to perceive depth. In this tests, seated participants wearing 3D glasses are shown images. Inability to see depth or in 3D will cause the images to appear as points instead of raised objects. The objects are presented in different stages, with each stage requiring participants to discriminate different levels of depth perception. The test is scored in optical units - ranging from 0 to 15 arc-seconds. The maximum score corresponds to the level where the last object was identified.
2. Convergence measured by "motor punctum proximum": (cm) When an object is moving towards our eyes, they symmetrically converge in order to maintain focus. There is, however, a point at which our eyes no longer symmetrically converge, which is referred to as the point of convergence or "motor punctum proximum". This test measures the distance (cm) between the bridge of the nose and the point of convergence in seated participants as an object is moved closer to their head.
3. Convergence fusional proximum: (diopters, prism convergence units) This test is similar to (2). When an object is moving closer to our head, our eyes symmetrically converge to maintain focus. However, when the object is moved beyond the participant's ability converge, the participant will begin to see two images (double vision). This test measures the distance between the bridge of the nose and the point where double vision (cm) occurs in seated participants as an object is moved closer to their head.
4. Binocular fusion with convergence: (diopters, prism convergence units) This test measures how well a participant can adapt to challenges in focusing light on the retina. This measure is comprised of two almost identical tests - differing only by distance. One test occurs when an object placed at 3m from the seated participant, and the other with an object placed at 30cm from the seated participant. Light from the object is passed through a prism - this is analogous to moving the object further from the body. In response, the eyes must diverge (separate) to focus on the object, just as they would if the image actually moved away from the body. Different prisms are used to create increasing challenges for the participants. The score for these tests is the maximum amount of prism convergence (dioptres, noted on the prism as one would note diopters on eye glasses) that the seated participant can accommodate at 3m and at 30cm.
5. Binocular fusion with divergence: (diopters, prism convergence units) This is the same test as (4), except that the prisms diverge the light and the participant has to converge (instead of diverge) their eyes to maintain focus. The score for these tests is the maximum amount of prism divergence (diopters, noted on the prism, as one would note diopters on eye glasses) that the seated participant can accommodate at 3m and at 30 cm.
6. Saccadic movements or oculomotor capacity: (Score = bad, medium, good) Saccadic movements are rapid movements of the eyes that abruptly alter the point of fixation. During this test, lights will appear and disappear - in different locations on the screen - at a rate of 100 flashes per minute, for a total of 2 minutes. The participant assumes a tandem stance (dominant foot placed in front of non-dominant foot and in line) and stands an arm's length away from the screen. The participant is told to keep his/her head still, only moving his/her eyes to focus on the appearing lights. The test result is scored by the clinician based on a global qualitative impression over the entire 2 minute duration of the tests, with 3 separate sub-scores on an ordinal scale for quality - for synchronization (bad, medium, good) and saccadic correction (many corrections, few corrections, no corrections). The three sub-scores are combined into an overall score according to our industry partner's (Apexk) proprietary algorithm.
7. Anatomic oculomotor deviation: (diopters, prism convergence units) This test measures the natural deviation of the eyes (heterophobia) and also allows for the detection of strabismus. In strabismus, anatomic deviation is easily detected as the individual's eyes are misaligned, such that the individual's dominant eye is looking at the object of interest, but the "lazy/deviated" eye is not. In heterophobia, anatomic deviation is not visible to the naked eye; in fact, the deviation must be triggered by covering one eye at a time in sequence, to trigger the deviation. This measure is comprised of two identical tests, differing by distance: one occurs with an object placed 3m from the seated participant (far vision), and the other with an object placed 30cm from the seated participant (near vision). In this test, seated participants focus on an object. The clinician covers and uncovers the participant's eyes to trigger movements and uses a prism to cancel these movements. The prism that achieves this cancellation of movements is the measure of anatomic deviation. The score of the test is the rating of the prism that achieves the movement cancellation, for the object placed at 30cm and at 3m. Participants with strabismus are excluded from our study as strabismus is a contraindication to post-concussion visual training.

The main objective of this study is to evaluate the correlation between the change in symptoms and the change in the results of the binocular vision tests. There are at least three milestone timepoints for each participant: baseline (M1), significant improvement in symptoms (M2), and when the participant is asymptomatic with activity or 3 months post baseline testing (M3). Participants that do not have significant improvement at least 2 weeks post-M1 - will be measured at 2 weeks (M*) to determine if the visual tests of function have improved. These participants will also still be measured at M2 and M3 - for a total of 4 visits.

These milestones represent patient states: symptomatic, improved, resolution/end of study. For our primary analyses, any patient who does not improve significantly over 3 months would have measures at M1, M*, and M3 (end of study). Because they would not have improved in symptoms, including them in a correlation between changes in symptoms and changes in test results is not meaningful. Therefore, they will be excluded from the primary analyses and will be analyzed separately. This is because the investigators are still interested in knowing whether the test results can change in the absence of a change in symptoms. The first step is to assess if there is a correlation between the score on BVT and the participants' symptoms (Sx) at each time a milestone occurs. For clarity, the analysis is conducted from a dataset where each line of data is represented by: Participant, Time (M1, M2, M3), Symptom Score, and BVT Score. The overall statistical model is:

E [BVT] = β0 + β1*Sx + β2*M2 + β3*Sx*M2 + β4*M3 + β5*Sx*M3 + ε

Where M2=1 when the Sx and BVT are measured at M2 and is equal to 0 otherwise, M3=1 when the Sx and BVT are measured at M3 and is equal to 0 otherwise, and ε refers to a random effect variable that is used to account for repeated measures on the same participants. In this model, the coefficient β1 is the association between all of the participants' symptom scores and the BVTs. This is because M2=M3=0, so the terms to the right of β1*Sx all equal 0. In this model, testing if the time of measurement (i.e. M1, M2, or M3) affects the correlation is straightforward. If the correlation is the same at M2 as it is at M1, then the coefficient, β3, will be 0. Similarly, if the correlation is the same at M3 as it is at M1, then the coefficient, β5, will be 0. If both β3, and β5 are found to be close to zero, then the associations are independent of the milestone at which the data were collected and the analysis will be re-run with all the data together in a simplified analysis to increase the power of subgroup analyses.

Next, the association in change of BVT with change in Sx will be measured. For these analyses, the data to the relevant milestones will be restricted. The statistical models are:

E [BVT M2 - BVT M1 | M2=1, M1=1] = β0 + β6*(SxM2-SxM1) + ε E [BVT M3 - BVT M2 | M3=1, M2=1] = β0 + β7*(SxM3-SxM2) + ε where BVT M# refers to the BVT measured at milestone number = #, and SxM# refers to the symptom score measured at milestone number = #.

If the values of β6 and β7 are found to be similar, then the associations are, again, independent of the milestones at which the data were collected. As above, the analysis will be re-run with all the data together in a simplified analysis to increase the power of subgroup analyses.

The above equations can be used to assess the association in change of total symptom score to change in total BVT score, change in any one symptom score and change in any one BVT, and changes in subgroups of symptom scores and changes in subgroups of BVTs. Because a deficiency in a particular visual function would be expected to cause only certain symptoms and only affect certain BVTs, our primary analyses will be restricted to 5 comparisons, discussed in the outcome measure section.

Gross stereoscopic acuity and anatomic oculomotor deviation are tests that measure visual function that existed prior to the concussion, and are, therefore, not expected to correlate with any changes in symptoms. These tests are conducted as part of a general visual examination.

The following symptoms in the SCAT3 are not expected to correlate with any visual tests: pressure in the head, neck pain, sensitivity to noise, feeling slowed down, confusion, drowsiness, trouble falling asleep, more emotional, irritability, sadness, nervous or anxious.

The secondary analyses will include associations between the total symptom score and the total BVT score, and the associations between the scores for each symptom and the scores for each binocular vision measure separately. In addition, the investigators will explore associations within subgroups of the participants based on clinician impression if there are abnormalities in the visual system at the first visit (y/n), time between concussion and baseline testing (<14 days, 14-28 days, >28 days), past history of concussion (y/n), and past treatment for psychological condition (y/n).

As concussions are common, this study has the potential to contribute to improved management for the many patients suffering from dizziness and other symptoms following a concussion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 16 years or older
* Diagnosis of concussion by a medical doctor
* Participants must have concussion-related symptoms lasting at least 8 days, and no more than 70 days at the time of recruitment.

Exclusion Criteria:

* Participants with strabismus or a history of treated strabismus
* Head trauma other than a concussion (minor head injury)
* History of migraine or known neurologic disorders

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our target population is healthy adults aged 16 to 30 with concussion symptoms for at least 8 days and no more than 70 days.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the change in 5 of the 7 BVT and only concussion symptoms that affect those particular BVTs. | For each participant, there will be at least 3 milestone timepoints: M1, M2, M3. If the participant does not demonstrate significant improvement within 2 weeks, he/she will be evaluated at the 2-week mark (M*).
  The correlation will be evaluated from the estimated change in BVTs associated with an increase in the sum of the scores for several symptoms by one score as measured by the SCAT3.
  The correlations will be restricted to the following comparisons: (1) Convergence measured by "motor punctum proximum" versus sum of "headache, sensitivity to light, difficulty concentrating, difficulty remembering, fatigue, low energy", (2) Binocular fusion with convergence versus sum of "headache, sensitivity to light, feeling fog, don't feel right, difficulty concentrating, fatigue", (3) "Convergence fusional proximum" versus sum of "headache, blurred vision, sensitivity to light, difficulty concentrating, difficulty remembering, fatigue, feeling fog", and (4) Binocular fusion with divergence versus sum of "headache, blurred vision, sensitivity to light, fatigue".

SECONDARY OUTCOMES:
Associations between the total concussion symptom score and the total binocular vision test score | For each participant, there will be at least 3 milestone timepoints: M1, M2, M3. If the participant does not demonstrate significant improvement within 2 weeks, he/she will be evaluated at the 2-week mark (M*).
  The association between the total concussion symptom score and the total BVT score will be estimated from the coefficients (β) of the regression model.
Associations between the scores for each concussion symptom and the scores for each BVT | For each participant, there will be at least 3 milestone timepoints: M1, M2, M3. If the participant does not demonstrate significant improvement within 2 weeks, he/she will be evaluated at the 2-week mark (M*).
  The association between the total concussion symptom score and the total BVT score will be estimated from the coefficients (β) of the regression model.
Demographic variables as modifiers of the correlation between the results of the binocular vision tests and concussion symptoms. | Demographic information and medical history will be collected at the first visit.
  The coefficients (β) (as estimated from the linear regression model) of each individual test will be compared across subgroups stratified by sex, level of education, use of corrective lenses, past medical history (history of concussion, depression, anxiety, attention deficit (hyperactive) disorder, migraines, and eye injury), use of medications (grouped by drug classes).
Change in tests in the absence of a change in symptoms | For each participant, there will be at least 3 milestone timepoints: M1, M2, M3. If the participant does not demonstrate significant improvement within 2 weeks, he/she will be evaluated at the 2-week mark (M*).
  If there are participants who do not improve significantly, the primary analysis will be repeated on this select group of participants. Although there might not be significant improvement, there might still be some change in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Shrier, MD, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campos EC, Cipolli C. Binocularity and photophobia in intermittent exotropia. Percept Mot Skills. 1992 Jun;74(3 Pt 2):1168-70. doi: 10.2466/pms.1992.74.3c.1168. PMID 1501986
- [Result] Dikmen S, Machamer J, Fann JR, Temkin NR. Rates of symptom reporting following traumatic brain injury. J Int Neuropsychol Soc. 2010 May;16(3):401-11. doi: 10.1017/S1355617710000196. Epub 2010 Mar 1. PMID 20188017
- [Result] Kerr ZY, Register-Mihalik JK, Kroshus E, Baugh CM, Marshall SW. Motivations Associated With Nondisclosure of Self-Reported Concussions in Former Collegiate Athletes. Am J Sports Med. 2016 Jan;44(1):220-5. doi: 10.1177/0363546515612082. Epub 2015 Nov 18. PMID 26582799
- [Result] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Result] McCrory P, Meeuwisse WH, Aubry M, Cantu RC, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen R, Guskiewicz KM, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport: the 4th International Conference on Concussion in Sport, Zurich, November 2012. J Athl Train. 2013 Jul-Aug;48(4):554-75. doi: 10.4085/1062-6050-48.4.05. No abstract available. PMID 23855364
- [Result] Ventura RE, Balcer LJ, Galetta SL. The Concussion Toolbox: The Role of Vision in the Assessment of Concussion. Semin Neurol. 2015 Oct;35(5):599-606. doi: 10.1055/s-0035-1563567. Epub 2015 Oct 6. PMID 26444405